CLINICAL TRIAL: NCT03897712
Title: A Study to Evaluate the Safety and Effectiveness of a Silicone Hydrogel Custom Contact Lens
Brief Title: A Study to Evaluate the Safety and Effectiveness of a Silicone Hydrogel Custom Contact Lens When Compared to Alden Optical HP Sphere Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 886
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Results first posted 2022-10-26 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-09

CONDITIONS: Contact Lens Wear
Keywords: Soft Contact Lens; Soft Contact Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Custom Samfilcon B Contact Lenses (Experimental): Participants will wear Bausch + Lomb investigational custom samfilcon B contact lenses daily for 3 months. Participants will be provided with ReNu MultiPlus Lubricating and Rewetting Drops for use as needed during the study. Participants will store their worn study lenses in a lens case filled with Biotrue multi-purpose solution (MPS).
  Interventions: Device: Custom Samfilcon B Contact Lenses; Device: ReNu MultiPlus Lubricating and Rewetting Drops; Device: Biotrue Multi-Purpose Solution
- Alden Optical HP Sphere contact lenses (Placebo Comparator): Participants will wear Alden Optical HP Sphere contact lenses daily for 3 months. Participants will be provided with ReNu MultiPlus Lubricating and Rewetting Drops for use as needed during the study. Participants will store worn study lenses in a lens case filled with Biotrue MPS.
  Interventions: Device: Alden Optical HP Sphere Contact Lens; Device: ReNu MultiPlus Lubricating and Rewetting Drops; Device: Biotrue Multi-Purpose Solution

INTERVENTIONS:
Device: Custom Samfilcon B Contact Lenses — Contact lens
  Arms: Custom Samfilcon B Contact Lenses
Device: Alden Optical HP Sphere Contact Lens — Hioxifilcon D, 54% water, Alden Optical HP Sphere lens
  Other Names: Alden Optical® HP Sphere lens
  Arms: Alden Optical HP Sphere contact lenses
Device: ReNu MultiPlus Lubricating and Rewetting Drops — For use as needed during the study.
  Other Names: Bausch + Lomb ReNu MultiPlus® Lubricating and Rewetting Drops
Device: Biotrue Multi-Purpose Solution — For daily rinsing, cleaning, disinfecting, and storing their lenses in lens cases during the study.
  Other Names: Bausch + Lomb Biotrue® MPS

SUMMARY:
This study is to evaluate the safety and efficacy of Bausch + Lomb custom samfilcon B (test) lens compared to the hioxifilcon D, 54% water, Alden Optical HP Sphere (control) lens when worn by participants who wear soft contact lens on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to read, understand, and provide written informed consent on the institutional review board (IRB)-approved informed consent form (ICF) and provide authorization as appropriate for local privacy regulations.
* Participants must have clear central corneas and be free of any anterior segment disorders in each eye.
* Participants must be myopic, require contact lens correction from -1.00 diopter (D) to -6.00 D, and wear contact lenses in each eye.
* Participants must be correctable through spherocylindrical refraction to 47 letters (0.0 logMAR) or better (distance, high-contrast) in each eye.
* Participants must be able and willing to comply with all treatment and follow-up/study procedures.
* Participants must be adapted soft contact lens wearers and agree to wear their study lenses on a daily wear basis for approximately 3 months.

Exclusion Criteria:

* Participants participating in any drug or device clinical investigation within 2 weeks prior to entry into this study and/or during the period of study participation.
* Participants who are women of childbearing potential (those who are not surgically sterilized or postmenopausal), who are currently pregnant, plan to become pregnant during the study, or are breastfeeding.
* Participants who have worn gas permeable lenses in either eye within the last 30 days or who have worn polymethylmethacrylate lenses in either eye within the last 3 months.
* Participants with any systemic disease currently affecting ocular health or which, in the Investigator's opinion, may have an effect on ocular health in either eye during the course of the study.
* Participants using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Participants with an active ocular disease in either eye or who are using any ocular medication.
* Participants who currently wear monovision, multifocal, or toric contact lenses in either eye.
* Participants with an ocular astigmatism >1.00 D in either eye.
* Participants with anisometropia (spherical equivalent) >2.00 D.
* Participants with any Grade ≥2 finding in either eye during the slit lamp examination. Participants with corneal infiltrates in either eye, of any grade, are not eligible to participate in this study.
* Participants with any "present" finding during the slit lamp examination in either eye that, in the Investigator's judgment, interferes with contact lens wear.
* Participants with any scar or neovascularization within the central 6 millimeters (mm) of the cornea in either eye. Note: participants with minor peripheral corneal scarring (that does not extend into the central area), that in the Investigator's judgment, does not interfere with contact lens wear, are eligible to participate in this study.
* Participants who are aphakic in either eye.
* Participants who are amblyopic in either eye.
* Participants who have had any corneal surgery (for example, refractive surgery) in either eye.
* Participants who are allergic to any component in the study care products.
* Participants who meet any of the following criteria:

  1. The participant is an employee of the investigative site.
  2. The participant, or a member of the participant's household, is an ophthalmologist, an optometrist, an optician, or an ophthalmic assistant/technician.
  3. The participant, or a member of the participant's household, is an employee of a manufacturer of contact lenses or contact lens care products (for example, Alcon, Bausch + Lomb, Ciba Vision, CooperVision, or Johnson & Johnson).
  4. The participant, or a member of the participant's household, is an employee of a market research firm.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Varughese, Study Director — Bausch & Lomb Incorporated
Locations (7):
- United States (7):
  - Bausch Site 1, San Francisco, California
  - Bausch Site 2, Denver, Colorado
  - Bausch Site 3, Sarasota, Florida
  - Bausch Site 4, Pittsburg, Kansas
  - Bausch Site 5, Warrensburg, Missouri
  - Bausch Site 6, Vestal, New York
  - Bausch Site 7, New Berlin, Wisconsin

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Custom Samfilcon B Contact Lenses | Alden Optical HP Sphere Contact Lenses
Started | 56; 112 eyes | 28; 56 eyes
Completed | 46; 92 eyes | 25; 50 eyes
Not Completed | 10; 20 eyes | 3; 6 eyes

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Custom Samfilcon B Contact Lenses | Alden Optical HP Sphere Contact Lenses | Total
Number analyzed (Participants) | 56 | 28 | 84
Age, Continuous [Mean (Full Range); unit: years] | 31.8 [18 to 40] | 31.3 [19 to 40] | 31.5 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 18 | 52
  Male | 22 | 10 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 47 | 23 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Distance High-contrast logMAR Lens VA
Description: Monocular distance high-contrast logarithm of the minimum angle of resolution (logMAR) lens visual acuity (VA) will be assessed at Week 1, Month 1, Month 2, and Month. For each eye LogMAR will be averaged at Week 1, Month 1, Month 2, and Month 3 visits, resulting in 1 value of "All Study" logMAR lens VA per eye.
Time Frame: Month 3
Population: Randomized participants who attended 3-month visit and had no major protocol deviations.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Arm/Group | Custom Samfilcon B Contact Lenses | Alden Optical HP Sphere Contact Lenses
Number analyzed (Participants) | 46 | 21
Number analyzed (eyes) | 92 | 42
LogMAR | -0.057 (0.0582) | -0.059 (0.0590)

2. Secondary Outcome: Proportion Of Eyes With Grade >2 Slit Lamp Findings
Description: Graded slit lamp findings will be assessed at Month 3. Each eye will be classified with respect to having 1 or more observations with Grade >2 (Yes, No) at any visit.
  Criteria of each grade: 0=None, 1= Trace, 2= Mild, 3=Moderate, 4= Severe. Higher grades are worse outcomes.
Time Frame: Month 3
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Custom Samfilcon B Contact Lenses | Alden Optical HP Sphere Contact Lenses
Number analyzed (Participants) | 56 | 28
Number analyzed (eyes) | 112 | 56
eyes | 1 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Custom Samfilcon B Contact Lenses | Alden Optical HP Sphere Contact Lenses
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/28
Other Adverse Events (participants affected / at risk) | 0/56 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT03897712/Prot_SAP_000.pdf